CLINICAL TRIAL: NCT03207555
Title: Ibrutinib Monotherapy in Early Stage Chronic Lymphocytic Leukemia (CLL) Without IWCLL/NCI-WG 2008 Treatment Indications But With High-Risk Features for Disease Progression
Brief Title: Ibrutinib as Early Therapy in Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0039; NCI-2018-01121 (Registry Identifier: NCI CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Malignant Neoplasms Stated as Primary Lymphoid Haematopoietic; Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
Keywords: Malignant neoplasms stated as primary lymphoid haematopoietic; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Leukemia; SLL; Ibrutinib; PCI-32765; Imbruvica
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Participants take Ibrutinib by mouth 1 time every day for up to 2 years (24 cycles).
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — 420 mg by mouth once daily.
  Other Names: PCI-32765; Imbruvica

SUMMARY:
The standard approach to managing chronic lymphocytic leukemia (CLL) and small lymphocytic leukemia (SLL) is to wait until you have symptoms before treatment is given.

The goal of this clinical research study is to learn if providing earlier treatment for CLL or SLL with ibrutinib in patients who do not have symptoms will be more effective than waiting until symptoms develop.

This is an investigational study. Ibrutinib is FDA approved and commercially available for the treatment of patients with CLL or SLL. It is considered investigational to give ibrutinib to CLL and SLL patients before symptoms develop.

The study doctor can describe how the study drug is designed to work.

Up to 50 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take ibrutinib by mouth 1 time every day. Each dose should be taken with about 1 cup (8 ounces) of water.

If you miss a dose of ibrutinib, it can be taken as soon as possible on the same day. You should take your next dose as scheduled. If you forget to take a dose, do not take extra capsules on the next day to "make up" the missed dose.

You will be given standard drugs, such as allopurinol or valacyclovir, to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks. If you have side effects, your dose of ibrutinib may be lowered or temporarily stopped until you recover from the side effects.

Length of Treatment:

You may take ibrutinib for up to 2 years (24 cycles). If at the end of 2 years you are benefitting from ibrutinib and the study doctor thinks it is in your best interest to continue taking it, other treatment options will be discussed with you to allow you to continue to take ibrutinib.

You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Study Visits:

Each cycle is 28 days.

On Day 28 of Cycles 1-3 and then every 3 cycles after that until Cycle 24 (Cycles 6, 9, 12, and so on):

* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a physical exam.
* You will have an EKG.

On Day 28 of Cycles 1, 3, 6, 12, and 24, blood (about 3 tablespoons) will be drawn to test for genetic mutations related to the disease. At Months 3, 6, and 12, additional blood (about 8 teaspoons) will be drawn for immune system testing.

On Day 28 of Cycles 6, 12, 18 and 24, you will have CT, MRI or PET/CT scan to check the status of the disease. Depending on the results of the CT, MRI or PET/CT scans, you may not need to have these scans repeated. The doctor will discuss this with you.

On Day 28 of Cycles 6, 12 and 24, you will have a bone marrow biopsy to check the status of the disease.

If the doctor thinks it is needed or if the disease gets worse, some tests/procedures, such as physical exams and blood draws for routine tests, may be repeated more often.

Long-term follow-up:

Every 3 months, during a regularly scheduled clinic visit (if you are still receiving care at MD Anderson) or by phone (if you are receiving care outside of MD Anderson), you will be asked how you are doing, if you are still taking ibrutinib, and if you have any side effects. If called, this call should last about 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be age >/=18 years at the time of informed consent, understand and voluntarily sign an informed consent, and be able to comply with study procedures and follow-up examinations.
2. No treatment indication according to IWCLL/NCI-WG (International Working Group in Chronic Lymphocytic Leukemia/National Cancer Institute-Working Group) 2008 criteria
3. Estimated time to first treatment of 3 years or less according to MDACC nomogram
4. ECOG performance status of 0-2
5. Male and female subjects who agree to use both a highly effective method of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence , or sterilized partner) and a barrier method (eg., condoms, vaginal ring, sponge, etc) during the period of therapy and for 30 days after the last dose of study drug for females and 90 days for males. OR Female subjects who are of non-reproductive potential (ie, post-menopausal by history - no menses for >/=1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy)
6. Adequate hepatic and renal function as indicated by all of the following: Total bilirubin </=1.5 x institutional Upper Limit of Normal (ULN) except for patients with bilirubin elevation due to Gilbert's disease or of non-hepatic origin who will be allowed to participate, provided bilirubin is </=3 x institutional ULN; an ALT </=2.5 x ULN; and estimated creatinine clearance (CrCl) of > 30 mL/min, as calculated by the Cockcroft- Gault equation.
7. PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder).
8. Free of prior malignancies for 3 years with exception of patients diagnosed with basal cell or non-metastatic squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast, who are eligible even if they are currently treated or were treated and/or diagnosed in the past 3 years prior to study enrolment
9. Diagnosis of CLL/SLL that meets IWCLL diagnostic criteria

Exclusion Criteria:

1. Receipt of any prior therapy for CLL. Patients who have received "early intervention" with INVAC-1 vaccine against hTERT will be eligible provided all of the following exist: i) They had no response to the vaccine treatment (persistent CLL >1% in bone marrow). ii) ≥3 months have elapsed since the last dose of vaccine. iii) No residual toxicities attributable to the vaccine exist at the time of study enrollment. iv) The patient does not meet IWCLL criteria for requiring treatment.
2. Richter Transformation
3. Active malignancy requiring systemic therapy, other than CLL, with the exception of: adequately treated in situ carcinoma of the cervix uteri; adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
4. Systemic anticoagulation with warfarin or other Vitamin K antagonists
5. Active and uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP) requiring daily prednisone dose of >/=20 mg
6. Current and concurrent use of strong CYP3A4 inhibitors or inducers
7. Pregnant or breast-feeding females
8. Uncontrolled and active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
9. Any other severe concurrent disease, or history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that, in the investigator's opinion, may place the patient at undue risk to undergo therapy with ibrutinib
10. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
11. History of ischemic stroke within 6 months prior to enrollment
12. Evidence of bleeding diathesis or coagulopathy within 3 months (eg, von Willebrand's disease or hemophilia
13. Any history of symptomatic intracranial hemorrhage
14. Major surgical procedure with 4 weeks of first dose of study drug; open biopsy, or significant traumatic injury within 7 days prior to enrollment date; anticipation of need for major surgical procedure during the course of the study
15. Minor surgical procedures, fine needle aspirations or core biopsies within 3 days prior to enrollment date. Bone marrow aspiration and/or biopsy are allowed
16. Serious, non-healing wound, ulcer, or bone fracture
17. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
18. Active, uncontrolled infection
19. Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded
20. Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification (see Appendix L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Burger, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibrutinib
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Participants With Complete Remission (CR) at 24 Months
Description: Complete Remission (CR): Peripheral blood lymphocytes below 4 x 10^9/L (4000/ƒÝL), Absence of significant lymphadenopathy (lymph nodes >1.5 cm in diameter) by CT(or PET) examination of neck, thorax, abdomen and pelvis, No hepatomegaly or splenomegaly by physical examination (and CT/PET if assessment was abnormal before therapy or if physical exam is inconclusive), Absence of constitutional symptoms, Neutrophils more than 1.5 x 10^9/L (1500/ƒÝL) without need for exogenous growth factors, Platelets more than 100 x 10^9/L (100 000/ƒÝL) without need for exogenous growth factors, Hemoglobin more than 110 g/L (11.0 g/dL) without red blood cell transfusion or need for exogenous erythropoietin, Bone Marrow aspirate and biopsy, demonstrating at least normocellular for age, with less than 30% of nucleated cells being lymphocytes. Lymphoid nodules should be absent. If the bone marrow is hypocellular, a repeat determination should be made in 4 weeks or when peripheral blood counts have recovered.
Time Frame: Up to 24 months
Population: Of the 23 participants registered on-study, 18 participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 18
Participants | 3

2. Primary Outcome: Participants With Partial Remission (PR) at 24 Months
Description: Partial Remission (PR) at least one of criteria 1-3, and one or more of the features listed in number 4. 1. A decrease lymphocytes by 50% or more from the value before therapy. 2. Reduction in lymphadenopathy, defined by the following: - A decrease in lymph node size by 50% or more either in the sum products of up to 6 lymph nodes, or in the largest diameter of the enlarged lymph node(s) detected prior to therapy. - No increase in lymph node, and no new enlarged lymph node. In small lymph nodes (</=2 cm), an increase of less than 25% is not considered to be significant. 3. A reduction in enlargement of the spleen or liver by 50% or more. 4. The blood count should show one or more of the following results: - Neutrophils more than 1, without need for exogenous growth factors. - Platelet counts greater than 100 x10^9/L (100 000/ƒÝL) or 50% improvement over baseline without need for exogenous growth factors. - Hemoglobin greater than 11
Time Frame: Up to 24 months
Population: Of the 23 participants registered on-study, 18 participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 18
Participants | 15

3. Secondary Outcome: Progression-Free Survival (PFS) at 24 Months
Description: Time from date of treatment start until the date of progression or death from leukemia.
Time Frame: 24 months
Population: Of the 23 participants registered on-study, 18 participants were evaluable.
Measure: Median (Full Range); unit: Months
Arm/Group | Ibrutinib
Number analyzed (Participants) | 18
Months | NA [NA to NA] — The Progression Free Survival was not met below the level of detection

4. Secondary Outcome: Overall Response at 24 Months
Description: Overall Response is participants who achieve Complete Remission (CR) or Partial Remission (PR) at 24 months of treatment.
Time Frame: Up to 24 months
Population: Of the 23 participants registered on-study, 18 participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: through 24 months
Arm/Group | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=23)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=23)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 13 (16)
Chills (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Eye disorders - Other, specify (Eye disorders) | 3 (3)
Fatigue (General disorders) | 17 (17)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (4)
Headache (Nervous system disorders) | 5 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Vascular disorders) | 7 (11)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 5 (6)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 7 (8)
Malaise (General disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Palpitations (Cardiac disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 6 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 8 (9)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9 (15)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03207555/Prot_SAP_000.pdf